CLINICAL TRIAL: NCT02595775
Title: A Randomized Controlled Trial of an Audit and Feedback Report to Improve Colonoscopy Performance
Brief Title: A Trial of an Audit and Feedback Report to Improve Colonoscopy Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Cancer Care Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 477-2014
Record Dates: First submitted 2015-07-10; First posted 2015-11-03 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Polyps
Keywords: endoscopy measures; audit and feedback; quality improvement; randomized controlled trial; Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Round 1: Intervention arm (Experimental): Half of the endoscopists in Ontario will receive an individualized audit & feedback report.
  Individualized A/F report.
  Interventions: Other: Individualized A/F report
- Round 1: Control (No Intervention): Half of the endoscopists in Ontario will NOT receive an individualized audit & feedback report.
- Round 2: Month 12 (Other): All endoscopists in Ontario will receive an individualized audit & feedback report at month 12.
  Individualized A/F report
  Interventions: Other: Individualized A/F report
- Round 2: Poor performers (Other): In Round 2, selected 60 poorer performers will be randomly assigned to receive one of the following interventions at month 12:
  1. A/F report plus a high intensity intervention
  2. A/F report plus a low intensity intervention
  3. A/F report alone
  Interventions: Other: A/F report plus a high intensity intervention; Other: A/F report plus a low intensity intervention; Other: A/F report alone

INTERVENTIONS:
Other: Individualized A/F report — Individualized A/F report containing 9 colonoscopy quality measures.
  Arms: Round 1: Intervention arm; Round 2: Month 12
Other: A/F report plus a high intensity intervention — E.g. Master class in colonoscopy
  Arms: Round 2: Poor performers
Other: A/F report plus a low intensity intervention — E.g. Access to a video/presentation on good colonoscopy technique followed by a post presentation assessment.
  Arms: Round 2: Poor performers
Other: A/F report alone
  Arms: Round 2: Poor performers

SUMMARY:
This project aims to measure the impact of a physician report card (also called an audit & feedback report) on colonoscopy performance. Endoscopists in Ontario will be randomly assigned to either receive the endoscopist report card or to no feedback. Using Ontario health administrative data, the quality of colonoscopy will be compared between those who received the report card and those who do not. The investigators will also measure the effect of receiving endoscopist report card on colonoscopy performance amongst endoscopists who perform poorly at baseline compared to those who do not. Further, the acceptability of two educational interventions that aim to improve the quality of colonoscopy will be evaluated by conducting one-on-one interviews with select participants. This study is critical to ensure that Canadians have access to the highest quality colonoscopy possible.

ELIGIBILITY:
Inclusion Criteria:

* All practising endoscopists in Ontario who performed at least 5 colonoscopies in 2014

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 833 (Actual)
Dates: Start 2015-09; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Change in polypectomy rate from baseline | At month 12
  Measure change in polypectomy rate from baseline

SECONDARY OUTCOMES:
Additional outcome 1- Change in cecal intubation rate | At month 12
  Change in cecal intubation rate from baseline
Additional outcome 2 - Change in annual colonoscopy volume | At month 12
  Change in annual colonoscopy volume from baseline
Additional outcome 3 - Change in poor bowel preparation rate | At month 12
  Change in poor bowel preparation rate from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jill Tinmouth, MD, Principal Investigator — Sunnybrook Health Sciences Centre

REFERENCES:
- [Derived] Tinmouth J, Sutradhar R, Li Q, Patel J, Baxter NN, Llovet D, Paszat LF, Rabeneck L. A Pragmatic Randomized Controlled Trial of an Endoscopist Audit and Feedback Report for Colonoscopy. Am J Gastroenterol. 2021 Oct 1;116(10):2042-2051. doi: 10.14309/ajg.0000000000001498. PMID 34515669